CLINICAL TRIAL: NCT03012763
Title: Pharmacokinetics of Sulfasalazine, Paracetamol, Fexofenadine and Valsartan After Oral Administration Using 240 ml Non-caloric Water, a Carbohydrate Enriched Drink and Grapefruit Juice in Correlation to the Intestinal Availability of Water as Quantified by MRI-based Volumetry in 9 Healthy Male and Female Subjects
Brief Title: Oral Pharmacokinetics of Sulfasalazine, Paracetamol, Fexofenadine and Valsartan Using Different Administration Mediums
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GIT-Physiol_2016
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Pharmacokinetics; Magnetic Resonance Imaging; Administration, Oral
MeSH Terms: interventions — Acetaminophen; Sulfasalazine; fexofenadine; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- non-caloric water (Placebo Comparator): 50 mg sulfasalazine given in 240 ml table water after 6 h fasting and 250 mg paracetamol, 120 mg fexofenadine and 40 mg valsartan given in 240 ml non-caloric water 3 h thereafter
  Interventions: Drug: Paracetamol; Drug: Sulfasalazine; Drug: Fexofenadine; Drug: Valsartan; Device: non-caloric water
- caloric drink (Active Comparator): 50 mg sulfasalazine given in 240 ml table water after 6 h fasting and 250 mg paracetamol, 120 mg fexofenadine and 40 mg valsartan given in 240 ml caloric drink 3 h thereafter
  Interventions: Drug: Paracetamol; Drug: Sulfasalazine; Drug: Fexofenadine; Drug: Valsartan; Device: caloric drink
- grapefruit juice (Active Comparator): 50 mg sulfasalazine given in 240 ml table water after 6 h fasting and 250 mg paracetamol, 120 mg fexofenadine and 40 mg valsartan given in 240 ml grapefruit juice 3 h thereafter
  Interventions: Drug: Paracetamol; Drug: Sulfasalazine; Drug: Fexofenadine; Drug: Valsartan; Device: grapefruit juice

INTERVENTIONS:
Drug: Paracetamol — Oral administration of 250 mg paracetamol
Drug: Sulfasalazine — Oral administration of 50 mg sulfasalazine
Drug: Fexofenadine — Oral administration of 120 mg fexofenadine
Drug: Valsartan — Oral administration of 40 mg valsartan
Device: non-caloric water — Oral administration of 240 ml non-caloric water
  Arms: non-caloric water
Device: caloric drink — Oral administration of 240 ml caloric drink
  Arms: caloric drink
Device: grapefruit juice — Oral administration of 240 ml grapefruit juice
  Arms: grapefruit juice

SUMMARY:
The purpose of this study is to determine pharmacokinetics of the probe-drugs sulfasalazine, given in 240 ml non-caloric water and paracetamol, fexofenadine and valsartan after oral administration, given in 240 ml non-caloric water, in 240 ml caloric drink or in 240 ml grapefruit juice prior to ingestion and to visualize the localization and to measure the filling volume of stomach, small intestine as well as ascending, transverse and descending colon by T2-weighted magnetic resonance imaging after oral administration of 240 ml water (non-caloric water), after administration of 240 ml caloric drink and after administration of 240 ml grapefruit juice.

ELIGIBILITY:
Inclusion Criteria:

* ethnic origin: Caucasian
* body mass index: ≥ 18.5 kg/m² and ≤ 30 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent

Exclusion Criteria:

* weight less than 45 kg
* claustrophobia
* tinnitus
* cardiac pacemakers, metallic, plastic or silicone implants, dental retainer or metal-containing tattoos and piercings, Permanent Make-Ups, intrauterine devices
* known allergic reactions/ hypersensitivity to the active ingredients used or to constituents of the study medication (e.g. lactose, lecithin, sulfonamides, salicylates)
* bronchial asthma (all stages) and other known allergic diseases
* existing cardiac, haematopoietic or hematological diseases and/or pathological findings, which might interfere with the drug's safety, tolerability and/or pharmacokinetics or the requirements for the magnetic resonance tomography
* known hyperkalemia, hyponatremia or hypovolemia or medications that may cause these conditions.
* Hepatic, renal or metabolic diseases and/or pathological findings, which might interfere with pharmacokinetics and pharmacodynamics of the study medication (e.g. liver failure, kidney failure, acute intermittent porphyria).
* gastrointestinal diseases and/or pathological findings, which might interfere with gastrointestinal motility and emptying processes and interfering with pharmacokinetics and pharmacodynamics of the study medication (e.g. ileus)
* Erythema exsudativum multiforme.
* Glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency).
* Acute, chronic or recurrent infections.
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* positive results in HIV, hepatitis B virus and hepatitis C virus screenings
* subjects who are on a diet which could affect gastrointestinal motility or the pharmacokinetics of the drug (vegetarian, vegan)
* eating disorders e.g. anorexia, bulimia
* heavy tea or coffee drinkers (more than 1l per day)
* lactation and/or pregnancy test positive or not performed
* subjects suspected or known not to follow instructions
* subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* subjects liable to orthostatic dysregulation, fainting or blackouts
* participation in a clinical trial during the last 3 months prior to the planned start of the study less than 3 months after last blood donation
* therapy with transdermal patches
* any systemically available medication within 2 weeks prior to the intended first administration unless because of the terminal elimination half-life complete elimination from the body can be assumed for the drug and/or its primary metabolites (except oral contraceptives)
* intake of grapefruit or poppy seeds containing products within 14 days prior to the start of the study
* Females who don't fulfil the criteria for contraception as listed in section 7.5.1 of this protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
area under the concentration time curve (AUC) | up to 51 h after drug administration
  Computed with the measured concentration of Paracetamol, Fexofenadine and Valsartan in blood samples.
area under the curve of small bowel water volume | up to 6.75 h after drug administration
  Dynamic enhanced magnetic resonance examination gradient-echo T2-weighted HASTE images (TR 1300 ms, TR 321 ms, flip-angle 160°) will be acquired on a 1.5 Tesla MRI. A tube filled with 20 ml water will be fitted on the abdomen of the volunteers in order to have an internal reference for imaging. The obtained MRI files will be investigated with common radiological software (OsiriX, Voxar 3D, Fiji, 3D slicer). From the DICOM files there will obtained: Gastrointestinal volumes and their kinetics for stomach, small bowel, colon segments and gallbladder.
gastric emptying rate | up to 6.75 h after drug administration
  Dynamic enhanced magnetic resonance examination gradient-echo T2-weighted HASTE images (TR 1300 ms, TR 321 ms, flip-angle 160°) will be acquired on a 1.5 Tesla MRI. A tube filled with 20 ml water will be fitted on the abdomen of the volunteers in order to have an internal reference for imaging. The obtained MRI files will be investigated with common radiological software (OsiriX, Voxar 3D, Fiji, 3D slicer). From the DICOM files there will obtained: Gastrointestinal volumes and their kinetics for stomach, small bowel, colon segments and gallbladder. Gastric emptying rate will be estimated as the half life of water volumen in the stomach.
lag-Time of sulfapyridine (orocecal transit times) | up to 51 h after drug administration
  Estimated as the first significant concentration (>50 or 100 ng/ml) of sulfapyridine in blood samples after administration of Sulfasalazine.

IPD SHARING:
Plan to Share IPD: No